CLINICAL TRIAL: NCT06836895
Title: The Effect of Combined High Intensity Interval Training and Inspiratory Muscle Training on Pulmonary Function and Exercise Capacity in COPD Patients
Brief Title: High Intensity Interval Training and Inspiratory Muscle Training
Acronym: training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Ahmad Saied Mohammad, Dr, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COPD
Record Dates: First submitted 2025-02-09; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Walking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study (Experimental): The study group (n=50) underwent 8 weeks combined HIIT and IMT. The HIIT protocol involved four intervals, each lasting 4 minutes, beginning at 70% of maximum power and building to a target intensity of at least 85% HRmax. The IMT sessions included 2-3 sets of 30 breaths (totaling 60-90 breaths per session), with a two-minute rest between sets, three days per week starting with 30% of PImax and reaching 60% of PImax.
  Interventions: Behavioral: HIIT and IMT
- control (Experimental): therapeutic education and self-based walking for 30 minutes
  Interventions: Other: walking

INTERVENTIONS:
Behavioral: HIIT and IMT — The HIIT protocol involved four intervals, each lasting 4 minutes, beginning at 70% of maximum power and building to a target intensity of at least 85% HRmax. The IMT sessions included 2-3 sets of 30 breaths (totaling 60-90 breaths per session), with a two-minute rest between sets, three days per week starting with 30% of PImax and reaching 60% of PImax.
  Arms: study
Other: walking — 30-min walking
  Arms: control

SUMMARY:
The goal of this clinical trial is to investigate the effect of combined high intensity interval training (HIIT) and inspiratory muscle training (IMT) on pulmonary function and exercise capacity in patients COPD. one hundred patients with COPD (GOLD II and III) with ages between 40 and 70 years participated in this study. The main question it aims to answer is whether combined high intensity interval training (HIIT) and inspiratory muscle training (IMT) have effect on pulmonary function and exercise capacity Pulmonary function tests, incremental cycle ergometer tests, 6 min walk tests and inspiratory muscle strength were performed and dyspnea and Health-related quality of life (HRQoL) were assessed before and after the intervention period.

DETAILED DESCRIPTION:
METHODS Study Design This study was performed as a randomized, controlled trial over 8 weeks and included two groups. The study procedures were carried out in the Department of Rehabilitation and Health Sciences, Prince Sattam Bin Abdulaziz University, Al-Kharj, Saudi Arabia between June 2024 and October 2024 Ethical consideration The study protocol was approved by the Standing Committee of Bioethics Research in Prince Sattam bin Abdulaziz University, Saudi Arabia (ID: SCBR-359/2024). The study was conducted in line with the principles of the Declaration of Helsinki. All study participants have signed a written informed consent form. The aim, procedures and potential risks of the study were explained to the study population.

Randomization A researcher, uninvolved in any other aspect of this study, conducted randomization by creating a block randomization schedule without stratifications. Initially, randomization codes were generated using Microsoft Excel (Microsoft Corporation, Redmond, WA). The allocation was then concealed in sequentially numbered, sealed, non-transparent envelopes. Eligible participants were subsequently directed to a researcher responsible for overseeing treatment, who assigned them randomly to either the study or control group.

Subjects:

A total of 144 clinically stable patients with COPD were recruited from local health facilities and nearby hospitals and clinics through advertisements to participate in this study and 100 completed the study follow-up.

The inclusion criteria were: 1) diagnosis of mild-to-severe COPD according to guidelines criteria with mild or severe airflow obstruction (GOLD II and III) (20), 2) Age ≥40 but ≤70 years.

COPD is defined by non-fully reversible airflow obstruction FEV1-FVC ratio less than 70% of predicted, FEV1 equal or more than 30% of predicted after bronchodilation. 3) Body mass index between 18 kg/m2 and <30 kg/m2, Exclusion criteria were: 1) any musculoskeletal, cardiovascular, or neurologic diseases that prohibited participating in HIIT, 2) Exacerbation of COPD, 3) Participation in a pulmonary rehabilitation program or organized exercise training in the last 6 months.

A specialized physician examined all participants to exclude those who did not meet the inclusion criteria and to ensure their safety for participation in a high-intensity exercise program. Written informed consent was obtained from each participant after an introductory session explaining the detailed evaluation and training procedures used in the study. All participants were instructed to maintain their regular physical activity and medications throughout the study period. Participants were assessed both at baseline and following the exercise intervention. Baseline demographics are presented in the left panel of Table 1.

Eligible subjects were randomly assigned to one of two groups either the exercise group (Ex group) practiced HIIT and IMT or the control group who received a program of therapeutic education and 30-min self-based cycling or walking on cycle ergometers or on treadmills. Pulmonary function tests, incremental cycle ergometer tests, cardiopulmonary exercise tests with gas exchange analysis, 6 min walk tests and inspiratory muscle strength were performed and Health-related quality of life (HRQoL) was assessed before and after the intervention period.

Sample size calculation The sample size was determined based on an estimated effect size (d = 0.65), derived from changes in PImax observed in Larson's study (21). To reject the null hypothesis, the probability was set at 0.05, with a power of analysis at 90%, calculated using G*power 3.1.9.7 software (University of Dusseldorf, Dusseldorf, Germany). A total of 100 participants were initially recruited. However, the sample size was increased to 120 to account for an anticipated dropout rate of up to 20%.

Anthropometrics assessments:

All participants were assessed for body weight and height. A weight and height scale (Detecto, made in USA) was used. Body mass index (BMI) was calculated using the following formula:

BMI = weight (kg) / height (m)2

Pulmonary function tests Lung function test was carried out by the same experienced personnel using Master Screen Body® Jaeger-Carefusion spirometer (22745 Savi Ranch Parkway, Yorba Linda, CA, USA). The test was repeated until three acceptable spirograms were obtained. A spirogram was considered acceptable if it was artifact-free, demonstrated adequate expiration, had a 6-second plateau at the end of the forced expiratory phase, and showed proper patient compliance. Measurements included FEV1, forced vital capacity, total lung capacity, and residual volume (22).

The diffusing capacity of the lung for carbon monoxide (DLco) was measured using the single-breath technique with Master Screen Body® Jaeger-Carefusion spirometer (22745 Savi Ranch Parkway, Yorba Linda, CA, USA) (23). Lung function parameters were determined as percentage of predicted according to participant's height, age and sex based on summary equations (24,25).

Exercise capacity An incremental cycle ergometer test on an upright cycle ergometer (Kettler ErgoRace, Virginia Beach, VA)) with continuous ECG-registration was conducted to measure peak workload (W peak). Patients began pedaling at an initial load of 20W, with the resistance increasing by 10W each minute until they reached exhaustion. During the exercise heart rate and breathing frequency were recorded every minute. Systolic blood pressure, perceived exertion (Borg RPE scale), and dyspnea (Borg CR-10 scale) were assessed every two minutes. All variables were also measured before exercise and at 1, 2, 4, and 10 minutes post-exercise.

Maximal incremental cardiopulmonary exercise testing (CPET) with continuous ECG monitoring was performed for the assessment of patients' exercise capacity using a Quark CPET metabolic cart (Cosmed, Rome, Italy) on a stationary cycle ergometer (800S, Ergoline, Bitz, Germany) according to the ATS guidelines (26).

The test started with a warm-up period without resistance lasting 5 min by pedaling at 20W then the load was increased by 10W every minute until exhaustion. CPET was terminated when patients indicated they had reached maximal effort due to muscle fatigue or dyspnea. The criteria for test termination included an inability to maintain a pedaling cadence (<60 rpm) combined with subjective signs of fatigue, such as sweating and hyperpnea and one or more of the following: peak VO2 greater than 80% of the predicted value, maximum heart rate exceeding 80% of the predicted heart rate, respiratory exchange ratio (RER) over 1.0, or reaching a VO₂ plateau (where oxygen uptake no longer increased despite a continuous rise in workload) (27,28). The measured cardiorespiratory parameters were heart rate, breathing frequency, minute ventilation, peak O2 consumption, minute ventilation, pulmonary oxygen uptake (VO2), carbon dioxide flow rejected by the ventilation system (VCO2), anaerobic threshold, and respiratory exchange ratio (RER). Systolic blood pressure, along with subjective ratings of perceived exertion (using the Borg RPE scale) and dyspnea (using the Borg CR-10 scale), were recorded every two minutes (29).

Functional exercise capacity Functional exercise capacity was assessed using the 6MWT conducted on a 30 m along a flat corridor according to the American Thoracic Society guidelines (30). Heart rate, respiratory rate, oxygen saturation, and dyspnea were assessed before and after testing. Each patient received standardized pre-test instructions and verbal encouragement every minute during the test. Two tests were conducted, with the first serving as a familiarization trial and not included in the analysis (31).

Respiratory muscle strength Respiratory muscle strength was evaluated by measuring PImax with a digital mouth pressure meter (Micro RPM®, Micro Medical, United Kingdom). The highest value from three trials-each varying by less than 10%-was recorded, with at least 30 seconds of rest between each attempt. A PImax of 60 cm H2O was set as the lower limit for normal (32).

Health-related quality of life Health-related quality of life (HRQoL) was assessed using the St. George's Respiratory Questionnaire (SGRQ) (33), is a standardized self-administered questionnaire designed to measure self-perceived health impairments and quality of life in individuals with airway diseases. It evaluates three domains-symptoms, activity limitations, and disease impact having 50 items with 76 weighted responses, including symptoms (eight items), activity (16 items), and impacts (26 items). The total score of the questionnaire, is rated from 0 to 100, where 0 represents the best quality of life and 100 represents the poorest quality of life.

COPD assessment test Participants' symptoms will be documented using the COPD Assessment Test (CAT) (34), an eight-item questionnaire covering topics such as cough, sputum production, chest tightness, breathlessness on hills or stairs, limitations in home activities, sleep quality, and fatigue. A higher score reflects a greater impact of COPD on the participant's life (35).

Dyspnea The modified Medical Research Council Dyspnea Scale (mMRC) was used to evaluate the severity of dyspnea. It is a 0-4 scale designed to measure the impact of dyspnea on physical activity in individuals with respiratory conditions. On this scale, a score of 0 indicates dyspnea only during intense physical exertion, while a score of 4 reflects severe breathlessness that prevents the individual from leaving the house or causes difficulty during activities such as dressing or undressing. Subjects are required to mark the level of activity at which they experience dyspnea (36).

HIIT protocols The exercise training was carried out on an outpatient basis for 8 weeks, with each session starting and ending with 10 minutes of cycling on an ergometer at 30%-40% of baseline peak power (WRpeak) for warm-up and cool-down. The high-intensity interval training (HIIT) protocol involved four intervals, each lasting 4 minutes, beginning at 70% of maximum power (WRpeak) and building to a target intensity of at least 85% of maximum heart rate (HRmax). Each interval was followed by a 3-minute active recovery period at 30% of WRpeak. The full interval block lasted 28 minutes, and the entire session was 42 minutes. Heart rate was continuously monitored with a Polar heart rate monitor (Polar V800, Polar Electro Oy, Kempele, Finland). All exercise sessions were supervised, with verbal encouragement given during intervals. Heart rate and Borg scale ratings were recorded at the end of each interval, aiming for approximately 90% of maximum predicted heart rate and a Borg rating of 5-7 on the modified Borg scale. During the 3-minute active rest phases, intensity was reduced to achieve a target heart rate of 50-60% of the predicted maximum. A respiratory physiotherapist supervised each session, providing guidance, encouragement, and ensuring safety (29).

IMT Prior to beginning IMT, study participants were provided with an overview of IMT by a trained physiotherapist. The maximum inspiratory pressure (PImax) was recorded before starting the training. All sessions were held at the same location and time of day in a well-ventilated room. Before each session, participants sat comfortably in a chair, and several parameters-including heart rate (HR), oxygen saturation (SpO2), systolic blood pressure (SBP), diastolic blood pressure (DBP), and Borg scale score-were measured. Once clinical stability was confirmed, subjects rested for a minimum of five minutes and began the session when they felt ready.

Participants sat in a relaxed position with their upper chest, shoulders, and arms supported. A nose clip was applied, and they were instructed to take the mouthpiece, seal their lips tightly, inhale deeply and slowly to increase tidal volume, and then exhale completely with minimal effort. They were advised to maintain diaphragmatic breathing and to keep their shoulders and legs relaxed throughout. Symptoms such as dizziness, fatigue, and shortness of breath were monitored closely, and heart rate and SpO2 were tracked with a pulse oximeter. The IMT sessions used the Threshold IMT® device (Respironics New Jersey, Inc., USA) and included 2-3 sets of 30 breaths (totaling 60-90 breaths per session), with a two-minute rest between sets, three days per week. Initially, participants began with a resistance requiring 30% of their PImax for the first week. This load gradually increased by 10% weekly to reach 60% of their PImax by the end of the first month. Weekly PImax assessments were conducted to ensure appropriate load adjustments. IMT then continued at 60% of each participant's PImax, adjusted weekly based on the most recent PImax measurement. All respiratory muscle strength assessments were performed by the same trained physiotherapist to maintain consistency.

Control group Participants carried out a supervised program for 8 weeks, 3 days per week. The program included therapeutic education and 30-min self-based cycling or walking on cycle ergometers and on treadmills. After each session, Borg's perceived exertion was measured.

Statistical analysis Statistical analyses were conducted using SPSS software version 23 (Chicago, IL). All data were expressed as mean ± SD. The Shapiro-Wilk test was used to check if the continuous variables followed a normal distribution. An independent t-test was performed to confirm the homogeneity of basic characteristics of parametric data between the two groups. A two-way mixed analysis of variance (ANOVA) (2 X 2, group x time) was used to explore the differences before and after treatment in the variables of interest between the HIIT and control groups. The p-value was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria

* diagnosis of mild-to-severe COPD according to guidelines criteria with mild or severe airflow obstruction (GOLD II and III)
* Age ≥40 but ≤70 years.
* Body mass index between 18 kg/m2 and <30 kg/m2,

Exclusion Criteria:

* any musculoskeletal, cardiovascular, or neurologic diseases that prohibited participating in HIIT,
* Exacerbation of COPD,
* Participation in a pulmonary rehabilitation program or organized exercise training in the last 6 months.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Pulmonary function tests (FEV1, FVC, TLC, IC, FRC, RV) in liter | 8 weeks
  Lung function test was carried out by the same experienced personnel using Master Screen Body® Jaeger-Carefusion spirometer (22745 Savi Ranch Parkway, Yorba Linda, CA, USA). The test was repeated until three acceptable spirograms were obtained. A spirogram was considered acceptable if it was artifact-free, demonstrated adequate expiration, had a 6-second plateau at the end of the forced expiratory phase, and showed proper patient compliance. Measurements included FEV1, forced vital capacity, total lung capacity, and residual volume (22).
Pulmonary function test (FEV1/FVC, RV/ TLC, DLCO, SpO2rest) in percentage | 8 weeks
  Lung function test was carried out by the same experienced personnel using Master Screen Body® Jaeger-Carefusion spirometer (22745 Savi Ranch Parkway, Yorba Linda, CA, USA). The pulmonary function test procedures were conducted repeatedly until three satisfactory spirograms were obtained. A spirogram was considered acceptable if it was artifact-free, demonstrated adequate expiration, exhibited final forced expiratory phase plateau lasting 6 seconds, and reflected proper patient cooperation. Measurements of forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), total lung capacity (TLC), and residual volume (RV) were taken (22). The single-breath technique was implemented to measure the diffusing capacity of the lung for carbon monoxide (DLco) using Master Screen Body® Jaeger-Carefusion spirometer (22745 Savi Ranch Parkway, Yorba Linda, CA, USA) (23). The pulmonary function parameters were recorded as absolute values and percentage of predicted according to participa
Pulmonary function tests (PaO2rest, PaCO2rest) in mmHg | 8 weeks
  Lung function test was carried out by the same experienced personnel using Master Screen Body® Jaeger-Carefusion spirometer (22745 Savi Ranch Parkway, Yorba Linda, CA, USA). The pulmonary function test procedures were conducted repeatedly until three satisfactory spirograms were obtained. A spirogram was considered acceptable if it was artifact-free, demonstrated adequate expiration, exhibited final forced expiratory phase plateau lasting 6 seconds, and reflected proper patient cooperation. Measurements of forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), total lung capacity (TLC), and residual volume (RV) were taken (22). The single-breath technique was implemented to measure the diffusing capacity of the lung for carbon monoxide (DLco) using Master Screen Body® Jaeger-Carefusion spirometer (22745 Savi Ranch Parkway, Yorba Linda, CA, USA) (23). The pulmonary function parameters were recorded as absolute values and percentage of predicted according to participa
Exercise capacity (peak workload (WRpeak) in watt | 8 weeks
  To measure peak workload (WRpeak), an incremental cycle ergometer test was conducted on a motorized cycle ergometer (Kettler ErgoRace, Virginia Beach, VA). Continuous ECG-registration was maintained throughout the test. The initial pedaling load was 20W, with the resistance increasing by 10W each minute until they reached exhaustion
Functional exercise capacity (six minute walk distance) in meters | 8 weeks
  The six minute walk test (6MWT) was used to evaluate the functional exercise capacity. A 30 m long flat corridor was used to conduct the test according to the American Thoracic Society guidelines (30). Assessment of heart rate, respiratory rate, oxygen saturation, and dyspnea were performed before and after testing. Before beginning the test, patients received instructions on the proper test procedures. Each patient was verbally encouraged every minute during the test. Patients performed the test twice, with the initial trial done to familiarize them with the test procedures and was not recorded (31).

SECONDARY OUTCOMES:
Health-related quality of life | 8 weeks
  Health-related quality of life (HRQoL) was assessed using the St. George's Respiratory Questionnaire (SGRQ) (33), is a standardized self-administered questionnaire designed to measure self-perceived health impairments and quality of life in individuals with airway diseases. It evaluates three domains-symptoms, activity limitations, and disease impact having 50 items with 76 weighted responses, including symptoms (eight items), activity (16 items), and impacts (26 items). The total score of the questionnaire, is rated from 0 to 100, where 0 represents the best quality of life and 100 represents the poorest quality of life.
Dyspnea | 8 weeks
  The modified Medical Research Council Dyspnea Scale (mMRC) was used to evaluate the severity of dyspnea. It is a 0-4 scale designed to measure the impact of dyspnea on physical activity in individuals with respiratory conditions. On this scale, a score of 0 indicates dyspnea only during intense physical exertion, while a score of 4 reflects severe breathlessness that prevents the individual from leaving the house or causes difficulty during activities such as dressing or undressing. Subjects are required to mark the level of activity at which they experience dyspnea (36).

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Sattam Binabdulaziz University, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No